CLINICAL TRIAL: NCT06362655
Title: ACTIBESE Project - Active Behaviour in School Education: Ecological Model Application on School Physical Education to Improve Active Behaviours in Schoolchildren. Cross-sectional and Intervention Study
Brief Title: ACTIBESE Project - Active Behaviour in School Education
Acronym: ACTIBESE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Carlos Cristi Montero, Fernando Rodriguez-Rodriguez, Pontificia Universidad Catolica de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANID/FONDECYT 2013/1230801
Record Dates: First submitted 2024-03-22; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity; Child Behavior; Family Support
Keywords: Physical activity; School-based intervention; Exercise; Health; Well-being
MeSH Terms: conditions — Sedentary Behavior; Child Behavior; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention Study
Masking Description: No apply
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIBESE Invervention Group (Experimental): Group that will receive the intervention from teachers to improve physical activity behaviors.
  Interventions: Behavioral: Intervention
- Traditional Physical Education Classes Group (Comparative group) (No Intervention): Group that won't receive the intervention from teachers for improving physical activity behaviours. This group will receive traditional physical education classes according to the national curriculum.

INTERVENTIONS:
Behavioral: Intervention — Intervention study. In this intervention study for teachers, a 5-month continuous training program will be included that will improve teaching style and promote teaching training. It will also strengthen teaching competencies to create teaching improvement strategies affecting PEaH and interpersonal and personal factors. This is expected to improve schoolchildren's AB, even when they are not directly influenced. The program will be designed according to the results of the cross-sectional study. The greatest associations found between the three proposed factors (school, interpersonal and personal factors) and schoolchildren AB will be sought. In addition, the characteristics of the schools and the possibilities of time and physical spaces available will be taken into account. This information will be recorded through validated questionnaires and interviews in the pre-test, post-test 1 and after follow-up post-test 2.
  Arms: ACTIBESE Invervention Group

SUMMARY:
The ACtive BEhaviour in School Education (ACTIBESE) project aims to assess and intervene in Chilean schoolchildren's active behaviours by examining the influence of personal, interpersonal, and school factors. This study includes a cross-sectional and intervention study involving 152 schools in the Valparaíso and Araucanía Regions, representing urban and rural areas. Participants, divided into children (8-11 years old) and adolescents (12-17 years old), will undergo a comprehensive evaluation, including sociodemographic characteristics, physical activity (PA) levels, parental and peer support, teaching styles of the teachers, and school environment characteristics.

For the cross-sectional study, questionnaires, interviews, accelerometry, and pedometry will be used to collect data on various factors influencing PA in schoolchildren. In the intervention study, a 5-month continuous training program for teachers will be implemented, focusing on improving teaching styles and enhancing teaching competencies related to physical education and health classes. The program aims to positively affect schoolchildren's PA indirectly through improved teaching practices.

The research will use mixed models, ANCOVA (Analysis of Covariance) , and logistic regressions for data analysis, incorporating multilevel logistic regressions to account for school-level dependencies. The study's outcomes will contribute valuable insights into the complex interactions between school, interpersonal, and personal factors influencing schoolchildren's PA, aiding the development of targeted interventions. This comprehensive approach aligns with the project's goal of fostering a physically active lifestyle among Chilean schoolchildren.

DETAILED DESCRIPTION:
ACTIve BEhaviour in School Education project (ACTIBESE) is a project funded by the National Agency for Research and Development (ANID) of the Chilean government (Code Nº: 1230801), which seeks to investigate and propose useful tools to increase levels of Physical Activity (PA) in schools. The project will consist of two parts: a cross-sectional study (first and second years) and an intervention study (third year), over a period of three years.

Recruitment

An invitation to participate will be sent to the principals of the participating schools. Once the schools agree to take part and are selected, a meeting will be held with both the representatives of the administrative management authorities and the schoolteachers to explain in detail the aims and stages of the project.

Subsequently, an informative meeting will be held with parents and schoolchildren using the same terms. The groups will be divided by age: children from grades 3-6 of primary school (8-11 years old) and adolescents from grade 7 of primary school to grade 2 of secondary school (12-16 years old).

Cross-sectional study

This study will determine the school factors associated with Active Behaviour (AB) in schoolchildren. These include teaching styles, teaching training, teacher perception of Physical Education (PE), and characteristics of the school and curriculum: school-environmental, spaces to play, infrastructure, recess, time dedicated and weekly frequency of PE, contents, topics, etc. This information will be obtained through qualitative questionnaires administered to schoolteachers. Additionally, the association between social factors and AB in schoolchildren will be studied. This will be determined through standardized questionnaires for parents. In addition, personal factors (i.e., motivation for PE, perception of PE, built-environment perception, and barriers to PA) will be evaluated using qualitative instruments (questionnaires). The outcomes of AB in schoolchildren will be evaluated using device-based methods (accelerometers and pedometers).

Intervention study

1. Assessment: This consists of applying the evaluation instruments to schoolteachers: Need-Supportive Teaching Style Scale (NSTSS), interviews, and focus group and schoolchildren: Young Activity Profile (YAP) questionnaire, "Pedalea y Anda al Cole" (PACO) questionnaire, accelerometry, pedometry, and barriers, both in the pre-test and post-test, to the intervention and control groups. In addition, instruments for parents (regarding interpersonal factors) will be used. The pre-test and post-test 1 correspond to the evaluation of the intervention process. Post-test 2 will evaluate the effect of the intervention through a follow-up process.
2. Intervention: The "teaching training" program consists of weekly class sessions addressed to teachers, where topics will be discussed to improve educational practices in Physical Education and Health (PEaH) classes, such as teaching strategies, teaching styles (productive style), recommendations for PA for children and the inclusion of the socioecological model, incorporating all the actors of the school educational environment. In addition, strategies are incorporated to stimulate the self-determination theory (SDT). This activity will be conducted in person; however, it will be changed to an online format according to the circumstances of the distance between cities. The "application of learning" will be carried out, where the teachers must apply the knowledge acquired in the teaching training to courses selected with a weekly frequency of one or two days. The application will take place over a semester (four months). To assess this implementation, pre-and post-tests will be carried out as defined in the methodology. Additionally, the teachers will keep a "field notebook" consisting of a record of the activities that go wrong or of complex situations that require a solution when the Teaching Training is applied in the chosen courses. Parallel to the problem, a solution or activity must be proposed to solve the difficulties that have arisen. Additionally, in the Teaching Training classes, teachers will be asked to attend various "workshops" on topics associated with AB and PEaH to diversify learning. To strengthen the process of applying these lessons, at least two mentoring sessions will be presented to the PEaH classes to resolve doubts, see the implementation of the changes, and understand the reality that schoolteachers face.

   This activity will be conducted in person; however, if the circumstances prohibit in-person meetings, it will be changed to an online format. In addition, regular "online meetings" will be established for schoolteachers to resolve questions and establish approaches, share ideas and concerns, and jointly resolve difficulties imposed on schoolwork or how to implement the different strategies learned in teaching training. This activity will take place every two weeks.
3. Follow-up: In this phase, teaching materials will be delivered to teachers to be applied during classes. In addition, there will be an observational follow-up to the process, a field notebook will be used, and two process evaluations will be conducted every six weeks from Post-test 1 through "mentoring." Additionally, a support web page will be created with help materials, and an app will be created for schoolteachers and schoolchildren to allow us to monitor the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least two PEaH classes per week, at least in selected grades.
* Grades between the 4th of primary and the 2nd of secondary .
* Each class had to include at least 15 schoolchildren.
* At least 15 informed consent forms per class for schoolchildren and 15 parents or guardians.
* At least two physical Education and Health (PEaH) schoolteachers.

Exclusion Criteria:

* No physical or mental disability
* Schoolteachers, schoolchildren, and parents cannot participate in other programs promoting physical activity (PA).

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels | 3 years
  Physical activity levels carried out inside school and outside school measured through the Young Activity Profile (YAP) questionnaire in the cross sectional stage and through the YAP questionnaire and accelerometry in the intervention stage.

CONTACTS AND LOCATIONS:
Locations (1):
- IRyS Group, School of Physical Education, Pontificia Universidad Católica de Valparaíso, Valparaíso, Chile., Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No